CLINICAL TRIAL: NCT02873858
Title: Elucidation of Sensory Characteristics and Food Preferences in the Elderly
Acronym: AUPALESENS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: PFITZENMEYER 2010
Record Dates: First submitted 2016-08-04; First posted 2016-08-22 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-07

CONDITIONS: Malnutrition
Keywords: elderly
MeSH Terms: conditions — Malnutrition | interventions — Smell

ARMS (4):
- 1.independent patients (Active Comparator)
  Interventions: Other: smell and taste tests
- 2. less mobile patients (Experimental)
  Interventions: Other: smell and taste tests
- patient in a residence (Experimental)
  Interventions: Other: smell and taste tests
- patients in a home for the elderly (EHPAD) (Experimental)
  Interventions: Other: smell and taste tests

INTERVENTIONS:
Other: smell and taste tests

SUMMARY:
Malnutrition is a frequent problem in persons older than 65 years: the prevalence of malnutrition can reach 25 to 29% in persons living at home who require help, figures vary between 19 and 38% for those living in institutions, and finally, the prevalence of malnutrition in hospitalized elderly patients can reach 30 to 90%. A few studies have attempted to explain modifications in attitudes, behaviour, the frequency of meals or nutritional status in the elderly by a fall in chemosensory sensitivity The aim of this project is to test the hypothesis that perhaps it is not as much the capacity to perceive a smell or a taste that affects eating behaviour in the elderly as their ability to distinguish between smells or tastes on the one hand (perceptual processing), and their ability to correctly interpret a chemosensory signal on the other (cognitive processing).

ELIGIBILITY:
Inclusion Criteria:

* Persons older than 65 years.
* Persons with diabetes, heart disease or hypertension stabilized by a treatment.
* Persons cognitively able to carry out the tests and fill in the questionnaires (Folstein test between 22 and 30).

Exclusion Criteria:

* Any person suffering from an acute disease at the time of the test.
* Any person presenting any allergy whatsoever (food, mites, pollen…).
* Any person suffering from asthma or severe respiratory disorders (lung cancer, tracheotomy…).
* Any person presenting anosmia (total loss of olfaction) from birth or following physical trauma (head injury) or due to disease (severe rhinitis).
* Persons with diabetes, heart disease or hypertension not stabilized by treatment.
* Any person presenting life expectancy of less than 6 months.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 611 (Actual)
Dates: Start 2010-12; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Indeed the level of dependency of scores at each of the olfactory tests, gustatory and masticatory | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France